CLINICAL TRIAL: NCT04571333
Title: Feasibility Study: A Totally Implantable Cochlear Implant (Mi2000) for Electrical Stimulation of the Auditory Pathway of Adults With Severe to Profound Sensorineural Hearing Loss
Brief Title: Feasibility of the Mi2000 Totally Implantable Cochlear Implant in Severely to Profoundly Deaf Adults.
Acronym: TICI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MED-EL_CRD_2014_03
Record Dates: First submitted 2020-09-09; First posted 2020-10-01 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Sensorineural Hearing Loss, Bilateral; Cochlear Implants
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mi2000 Cochlear Implant surgery (Experimental): During the surgery visit, the Mi2000 Cochlear Implant will be implanted according to the general surgical guidelines and the Mi2000 specific surgical guidelines under general anaesthesia.
  Interventions: Device: Mi2000 Totally Implantable Cochlear Implant

INTERVENTIONS:
Device: Mi2000 Totally Implantable Cochlear Implant — During the surgery visit, the Mi2000 Cochlear Implant will be implanted according to the general surgical guidelines and the Mi2000 specific surgical guidelines under general anaesthesia.

SUMMARY:
This clinical investigation aims to collect data on the use of the Mi2000 system, a totally implantable cochlear implant system, for the first time in human subjects.

DETAILED DESCRIPTION:
Cochlear implants (CI) provide a large majority of recipients with a significant degree of speech understanding. However, CI systems rely on external parts, namely Behind-the-Ear (BTE) audio processors with coils or single-unit processors to function. This can have several disadvantages: for instance, the hardware is exposed to external trauma and to the effects of head movement and gravity. The device is also put at risk by humid, dusty, or dirty conditions as well as by physical activities that lead to water exposure such as swimming or sports in general (e.g. perspiration).

In addition, some patients are concerned with the cosmetic appearance of the external parts which are visible (more so than modern behind-the-ear hearing aids), something that may not be desirable to many potential candidates.

This clinical investigation aims to collect data on the use of the Mi2000 system, a totally implantable cochlear implant system, for the first time in human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of eighteen (18) years at time of enrolment
* Bilateral sensorineural hearing loss with no or limited benefit from a hearing aid (>70 dB HL PTA4)
* Post-lingual onset of deafness
* No or limited benefit from hearing aids for less than 10 years.
* A maximum score of 50% on a monosyllables test in the language of the test centre in the ear to be implanted
* General health condition, psychological and emotional condition deemed compatible with the treatment and tests performed in this study and realistic expectations, as deemed appropriate by the implanting surgeon/implant board
* Fluency in the test language with excellent proficiency, as appropriate to perform speech testing
* Evidence of up-to-date vaccinations against meningitis, as per recommendations by the applicable national body
* Signed and dated informed consent before the start of any study-specific procedure

Exclusion Criteria:

* Lack of compliance with any inclusion criterion
* Previously having received an implant on the location chosen for placing the cochlear implant
* Having received a hearing implant from another manufacturer than MED-EL on the contralateral ear
* Pre-existing condition known to necessitate MRI scans after implantation of the Mi2000
* Women being pregnant or nursing
* Women of child-bearing age not reporting to use effective contraception
* Contraindication to surgery in the middle and inner ear
* Contraindication to general anaesthesia
* Cochlear malformations, ossification or other obliteration of the cochlea, history of meningitis preventing placement of the electrode array, as confirmed by medical examination
* Acute cholesteatoma
* Acute external or middle ear infections
* Perforated tympanic membrane
* Known intolerance to any of the materials used for the implant or accessories
* Non-functional auditory nerve and/or upper auditory pathway including a history of vestibular schwannoma
* Factors preventing appropriate placement of the stimulator housing and the microphone, including fixation with screws, in the bone of the skull
* Unstable Meniere's disease, Auditory Neuropathy, Epilepsy not responding to treatment
* Unrealistic expectations of the subject
* Permanent inability and/or unwillingness to participation in post-operative care and rehabilitation
* Known intellectual disability and/or psychological diseases
* Participation in other pharmacological clinical trials within four weeks prior to enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Safety of the study device | up to 16 weeks
  Safety of the study device in the intended population will be assessed by an analysis of adverse events (AEs) reported

SECONDARY OUTCOMES:
Safety of the study device | up to 52 weeks
  Safety of the study device in the intended population will be assessed by an analysis of adverse events (AEs) reported
Speech perception in quiet | up to 52 weeks
  Speech perception in quiet will be assessed with a monosyllables test
Speech perception in noise | up to 52 weeks
  Speech perception in noise will be assessed with a sentence test in noise
Audiograms | up to 52 weeks
  Audiograms will be recorded in unaided and in best aided condition
Impedance Field Telemetry | up to 52 weeks
  Impedance Field Telemetry (PIFT)
Auditory Nerve Response Telemetry (ART) | up to 52 weeks
  Auditory Nerve Response Telemetry (ART)
Hardware and device parameters stored in the internal memory | up to 52 weeks
  Readout of device parameters stored in the devices internal memory (e.g. log files, battery status, charging status, usage times)
Questionnaire on usability of the device | up to 52 weeks
  Device use will be assessed using a questionnaire, recording user feedback
Health Utilities Index 2/3 (HUI2/3) | up to 52 weeks
  Quality of life will be assessed by the HUI2/3 questionnaire
Speech, Spatial and Qualities of Hearing (12 item version) (SSQ12) | up to 52 weeks
  Quality of life will be assessed by hte SSQ12 questionnaire
Nijmegen Cochlear Implant Questionnaire (NCIQ) | up to 52 weeks
  Quality of life will be assessed by the NCIQ questionnaire
Sound quality ratings | up to 52 weeks
  Subjective rating of sound quality

CONTACTS AND LOCATIONS:
Overall Officials: Phillippe Lefebvre, Prof. Dr. med., Principal Investigator — Centre Hospitalier Universitaire de Liège, ORL; Joachim Müller, Prof. Dr. med., Principal Investigator — Klinikum der Universität München, HNO
Locations (2):
- Centre Hospitalier Universitaire de Liège, Department ORL, Liège, Belgium
- Klinikum der Universität München, Campus Großhadern, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Due to small sample size, de-identification of individual patient data is not possible.